CLINICAL TRIAL: NCT04955977
Title: Effects of a Physical Exercise Program on the Responses Measured by HIF-1 Related to Ventilatory and Hematological Function in Patients With COPD Resident at 2600 m.s.n.m.
Brief Title: Physical Exercise and Responses Measured by HIF-1 in COPD
Acronym: ECOPDHIF-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 47970
Record Dates: First submitted 2021-06-15; First posted 2021-07-09 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Exercise; Hypoxia; Epigenomics; Therapeutics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Hypoxia | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study with assignment to groups by convenience by severity of the disease. Group 1: COPD GOLD1-2, Group 2: COPD GOLD3-4, Group 3: Control. Study with intra- and inter-group comparison before and after intervention with an external control group
Who Masked: Participant
Masking Description: Unique masking when study participants, who will not know:
  1. Assignment to research groups, for which the measurement of the severity of the disease will be developed individually.
  2. Treatment to receive, for which the intervention will be carried out individually and at the home of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G1: People with a diagnosis of COPD stratified in GOLD 1-2. (Experimental): * Adult person, over 40 years of age, both sexes, resident in medium altitudes or 2,600 meters above sea level in the last 2 years.
  * People with a diagnosis of COPD categorized in GOLD 1-2, with no record of respiratory crises in the last 3 months.
  * People with a diagnosis of COPD categorized by lung function in GOLD 1,2,3 and 4 and by severity of symptoms in A, B and C, without the need for supplemental oxygen.
  * People with a diagnosis of COPD settled and domiciled for a minimum time of 14 months at moderate altitudes or 2600 m.a.s.l.
  * People who have read and signed informed consent and who have membership in a mandatory health plan.
  Interventions: Other: Physical exercise program; Other: Health education in COPD
- G2: People with a diagnosis of COPD stratified in GOLD 3-4. (Experimental): * Adult person, over 40 years of age, both sexes, resident in medium altitudes or 2,600 meters above sea level in the last 2 years.
  * People with a diagnosis of COPD categorized in GOLD 1,2,3 and 4, with no record of respiratory crises in the last 3 months.
  * People with a diagnosis of COPD categorized by lung function in GOLD 3-4 and by severity of symptoms in A, B and C, without the need for supplemental oxygen.
  * People with a diagnosis of COPD settled and domiciled for a minimum time of 14 months at moderate altitudes or 2600 m.a.s.l.
  * People who have read and signed informed consent and who have membership in a mandatory health plan.
  Interventions: Other: Physical exercise program; Other: Health education in COPD
- G3: Control - People without a COPD diagnosis. (Active Comparator): Healthy people, over 40 years old. No history of cigarette smoking or exposure to wood smoke. Who do not present diagnoses of musculoskeletal injuries and who are residents at 2600 meters above sea level for more than 14 months. With affiliation to a mandatory health plan and signature of informed consent.
  Interventions: Other: Physical exercise program

INTERVENTIONS:
Other: Physical exercise program — Step 1 • Diaphragmatic reeducation: • Aerobic capacity: Intensity: zone 2, 60% HRMax, 4-6 / 10 Borg Scale; Charge: 20 m.
  Step 2 • Aerobic capacity: Intensity: zone 2, 65% HRMax, 4-6 Borg Scale; Charge: 25 m. • Muscular strength: Method: Pyramidal; Intensity: 3-4 / 10 Omni-Res; Load: 20% 1RM; Series: 3; Reps: 1. • Flexibility and elasticity: Intensity: 31-60 Perflex Scale; Charge: 10 - 20 s.
  Step 3 • Aerobic capacity: Intensity: zone 3, 70% HRMax, 5-6 / 10 Borg scale, Load: 25 m. • Muscular strength: Method: Pyramidal; Intensity: 4-5 / 10 Omni-Res; Load: 30% 1RM; Series: 4; Reps: 10. • Flexibility and elasticity: Method: active stretching; Intensity: 31-60 Perflex Scale; Charge: 10 - 20 s.
  Step 4 •Aerobic capacity: Intensity: zone 3, 75% HRMax, 6-7 / 10 Borg scale, Load: 30 m. • Muscular strength: Intensity: 5-6 / 10 Omni-Res; Load: 40-50% 1RM; Series: 4 s; Reps: 13. • Flexibility and elasticity: Method: active stretching; Intensity: 31-60 Perflex Scale; Charge: 10 - 20 s.
  Other Names: Therapeutic exercise
Other: Health education in COPD — Week 1-2: Health education: COPD and respiratory care at home. Week 3-4: Importance of daily physical activity in COPD. Week 5-6: Early Signs of COPD Exacerbation and Action Plan Week 7-8: Use and care of respiratory devices at home.
  Other Names: Health education
  Arms: G1: People with a diagnosis of COPD stratified in GOLD 1-2.; G2: People with a diagnosis of COPD stratified in GOLD 3-4.

SUMMARY:
Despite being considered a potentially preventable disease, COPD is classified as one of the respiratory problems with the highest prevalence and socioeconomic impact. According to the Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD), people with COPD require actions that optimize quality of life by improving lung function and increasing tolerance to fatigue.

Research such as those carried out by Semenza, establish that metazoan organisms such as the human species present biomolecular mechanisms for O2 homeostasis, based on transcriptional changes that allow regulating or modifying the responses necessary for the maintenance of the cellular metabolic functions. Hypoxia Induced Factor 1 (HIF-1) is the primary molecular mechanism for the regulation of O2-regulated genes in nuclear cells; Therefore, they promote adaptive mechanisms to hypoxia, through the generation of protein synthesis that favor processes such as erythropoiesis, angiogenesis, changes in oxidative metabolism and modification of the pulmonary vascular response.

Research carried out in cells of people with COPD exposed to environmental hypoxia by low oxygen pressure (PO2), have shown changes in the nuclear concentrations of HIF-1, affecting the transcriptional mechanisms of specific genes for Erythropoietin (EPO), the Factor of Vascular Endothelial Growth (VEFG) and therefore limit the generation of essential proteins for systemic responses. These transcriptional mechanisms are conditioned by the structural changes of chromatin seconded by the inhibition in the performance of histone enzymes, which influences the synthesis of proteins involved in metabolic, hematological and / or ventilatory processes as a response. to hypoxia. However, the concentration and effect of HIF 1 on the synthesis of EPO and VEGF and its relationship with spirometric and hematological tests have not been studied in COPD people who live in medium altitudes and who are additionally exposed to additional hypoxic stimuli such as exercise physical.

Although it is known that in COPD there is a decrease in the diffusion of O2 through the blood-gas barrier generating hypoxia and that with low PO2 there are biomolecular adaptations to favor oxygenation, perfusion, and metabolism; At the moment, the responses of HIF-1 and its effect on the generation of proteins associated with erythropoiesis and angiogenesis (EPO, FEVG) in people with COPD with physical exercise-based treatments are unknown.

DETAILED DESCRIPTION:
1. General objective

   To determine the effect of a physical exercise program on the responses mediated by HIF-1 in COPD patients resident at 2600 m.s.n.n.
2. Research question.

   What is the effect of a physical exercise program on the responses mediated by HIF-1 in COPD patients resident at 2600 m.s.n.n?
3. Type of study.

   It is presented as a quasi-experimental study with intra- and inter-group comparison before and after, with an external control group. Two observations will be made in time (pre and post test); Comparisons will be made intra-group and between groups, as follows:

   Experimental group 1:
   * G1: People with a diagnosis of COPD stratified in GOLD 1-2.
   * O1: Measurement of HIF-1, HADC 7, EPO Synthesis, VGEF Synthesis, FEV1, Hemogram.
   * X: Application of the physical exercise program.
   * O2: Measurement HIF-1, HADC 7, EPO Synthesis, VGEF Synthesis, FEV1, Hemogram.

   Experimental group 2:
   * G2: People with a diagnosis of COPD stratified in GOLD 3-4.
   * O3: Measurement HIF-1, HADC 7, EPO Synthesis, VGEF Synthesis, FEV1, Hemogram.
   * X: Application of the physical exercise program.
   * O4: Measurement HIF-1, HADC 7, EPO Synthesis, VGEF Synthesis, FEV1, Hemogram.

   Control group:
   * G3: People without a COPD diagnosis.
   * O5: Measurement of HIF-1, HADC 7, EPO Synthesis, VGEF Synthesis, FEV1, Hemogram.
   * X: Application of the physical exercise program.
   * O6: Measurement HIF-1, HADC 7, EPO Synthesis, VGEF Synthesis, FEV1, Hemogram.
4. Phases of the study

   Phase 1. Enrollment of participants and identification of baselines of HIF-1 measurements, synthesis of VEGF and EPO, Spirometry and Hemogram. Phase 2. Piloting and application of the physical exercise program in COPD residents in medium altitudes. Phase 3. Final measurement of HIF-1, synthesis of VEGF and EPO, Spirometry and Hemogram; Phase 4. Analysis of intra and intergroup results, writing final research report, socialization and publication of results.

   The pilot test will be carried out with 10% of the initial sample calculated, in order to evaluate and refine the instruments to be used, verify the conditions of application of these and the procedures involved in obtaining the data, such as the times of registration of participants' participation in each session, execution of the physical exercise program and application of measurement tests.
5. Sample size.

   A sample size calculation will be performed for longitudinal studies, using the Diggle formula for both differences between individuals and between groups, taking as a reference an expected effect, differences of 7.1, 4.96, 1.14 and 0.19 for the HIF-1; 1.6, 1.1; and finally 0.6, 0.3, 0.23 and 0.052 for the effect on VEGF and EPO protein synthesis. Similarly, variances (δ2) between 0.00004489 to 6.76 were considered depending on each effect measure as reported in the literature, Table 3 shows the expected variances and effect magnitudes in detail. Additionally, two measurements (pre and post) will be considered, for one (n = 4) for three comparison groups, with a type I error of α = 0.05, power P = 0.80 and exploring correlations (ρ) between -0.86 , 0.4, 0.47, 0.6, 0.79 or 0.8 depending on each parameter.

   Below, you can see the different scenarios where the study sample is sufficient, it is thus that for the value of the expected effect magnitude in each of the response variables with the different scenarios of variances and correlations raised, the sample can be between 1 to 2630 participants. For the consideration of the present study, a sample of 27 participants will be taken in order to be able to observe different magnitudes with sufficient power. Because there may be losses to follow-up, a 20% increase was made for a total of 33 participants, 11 per group (66 total measurements).
6. Selection and enrollment of participants.

   After obtaining the endorsements of the research and ethics committees of the National University of Colombia, the study population will be called; This will be done in person and via telephone to potential participants of the research project. The call mechanism will be by: 1. Lists of people attending rehabilitation programs of hospital institutions, 2. Open invitation to possible participants, through radio calls, newspapers and social networks, 3. Direct invitation to known people who comply with the inclusion criteria. Once the invitation is made, a screening will be carried out to identify the inclusion and exclusion criteria; Next, an appointment will be scheduled with the participant to fill out the informed consent.
7. Evaluation of the health condition and assignment of study groups.

   People interested in participating in the research and who have signed informed consent, will be initially summoned for the medical and therapeutic evaluation of their health condition, therefore a clinical history format is presented for this project (Annex 3); At this time, spirometry will be applied to determine the degree of pulmonary compromise according to what is presented by the GOLD report 2019. Additionally, the physical fitness of the participants will be measured for the prescription of physical exercise.
8. Data analysis

   8.1. Descriptive analysis

   For the descriptive analysis of the characteristics of the population studied, the variables on the qualitative measurement scale will be described as proportional frequencies, the continuous variables will be described with measures of central tendency (mean and median) and dispersion (standard deviation, interquartile range). according to whether or not they present a normal distribution according to graphic (histograms, dispersion, among others) and numerical (Shapiro-Wilk) methods.

   8.2 Baseline analysis

   To compare the three groups (G1: COPD 1-2, G2: COPD 3-4, G3: without COPD). Parametric and non-parametric tests will be carried out according to the verification of a priori criteria. For comparisons between proportions, Chi2 or Fischer's exact will be carried out, for the comparison of continuous variables between the three groups an ANOVA or kruskal wallis test will be used.

   8.3 Multivariate analysis

   As a longitudinal method, a repeated measures analysis will be carried out for correlated data. For each of the continuous outcome variables, the analysis will be performed with fixed effects (marginal) models. The evaluation of the assumption of normal distribution of the variables will be carried out using graphic methods (histograms, box plots and QQ graphs).

   In the model, the main exposure will be included as covariates, referring to the group it belongs to (G1: COPD 1-2, G2: COPD 3-4, G3: without COPD). The time will be taken as a continuous variable according to the minutes between each of the measurements, for which its linearity and its interactions with the covariates of interest will be evaluated, in case of not complying with this assumption it will be categorized based on the measurements carried out, considering the baseline measurement as a reference and the evaluation of possible interaction terms will be carried out. For the variables with normal distribution, the restrictive model of maximum likelihood (REML) will be used to select the best correlation matrix; later, to select the covariates to keep in the model, the maximum likelihood estimate (MLE) will be used. The selection of the best model will be based on the lower value of the Akaike information criterion (AIC) and the Bayesian evaluation criterion (BIC) after having evaluated the interactions and the non-linear terms. For conditional models, models with intercept and slopes will be used. If it does not present a normal distribution, a generalized equation estimation model (GEE) with an unstructured matrix will be implemented. A residual analysis will be performed on all final models. With the above, it will be possible to evaluate the effects both within and between groups with a more robust model to analyze the outcome measures and control for possible confounding variables.
9. Intervention (Physical exercise program for people with COPD.)

   The physical exercise program is proposed according to the existing scientific evidence and the recommendations of the GOLD 2019. This program will be based on an 8-week macro training cycle with 3 sessions per week for a total of 24 out-of-hospital training sessions. It will consist of 4 steps, each one consisting of 2 training microcycles or 6 work sessions; Training of conditional and coordinative physical qualities will be carried out in each step, and additionally with health education sessions.
10. Control of biases

10.1. Control and management of internal invalidation sources

* Threat-History. Actions to be taken: Participants in the experimental groups experience the same event, being people with COPD exposed to altitude hypoxia due to being residents at 2060 meters above sea level, with stratification of disease severity (GOLD 3 - 4).
* Threat - Maturation. Actions to be taken: Establishment of inclusion and exclusion criteria. Participants over 40 years of age with complete biological maturation.
* Threat-Instability of the measuring instrument. Actions to be taken: The instruments to be used in the collection of information have validity and reliability; They have been used in multiple investigations related to the subject and are strategies.
* Threat-Instability of the experimental environment. Actions to be carried out: the environmental conditions are the same for all the research participants since they will be applied at 2,600 meters above sea level in the city of Bogotá D.C. The intervention has a defined protocol that will be applied by the same researcher to all study participants.
* Threat: Instrumentation. Actions to be taken: the same measurement instruments will be applied to all research participants regardless of the stratification of the disease or the assignment to the control group.
* Threat - Selection. Actions to be taken: Participants will be established in groups according to the GOLD 3 or GOLD 4 disease stratification.
* Threat-attrition. Actions to be taken: Calculation of the sufficient sample size and carried out by a statistician outside the investigation, taking into account 20% of possible attrition.

10.2 Control and management of sources of external invalidation

* Threat-Reactive or interaction effect of the tests. Actions to be taken: The instruments that will be used in the collection of information have validity and reliability.
* Threat-Effect of interaction between selection errors and experimental treatment. Actions to be taken: Inclusion and exclusion criteria are established, which rule out people with aspects that can be inferred from the research results.
* Threat-Interference from multiple treatments. Actions to be taken: A single physical exercise program will be carried out for all the research participants.
* Threat: Impossibility of replicating the treatments: Actions to be taken: Detailed description of the content of the physical exercise program.
* Threat-Interaction between history or place and the effects of the experimental treatment. Actions to be carried out: The investigation will be carried out in the same place and laboratory, located at 2,600 meters above sea level, in the city of Bogotá D.C.

ELIGIBILITY:
Inclusion Criteria:

* Adult person, over 40 years of age, both sexes, resident in medium altitudes or 2,600 meters above sea level in the last 2 years.
* People with a diagnosis of COPD categorized in GOLD 1,2,3 and 4, with no record of respiratory crises in the last 3 months.
* People with a diagnosis of COPD categorized by lung function in GOLD 1,2,3 and 4 and by severity of symptoms in A, B and C, without the need for supplemental oxygen.
* People with a diagnosis of COPD settled and domiciled for a minimum time of 14 months at moderate altitudes or 2600 m.a.s.l.
* People who have read and signed informed consent and who have membership in a mandatory health plan.

Exclusion Criteria:

* People with a medical diagnosis of anemia, liver disease, chronic kidney disease, rheumatological diseases or a history of gastrointestinal bleeding in the last 2 months.
* People with a diagnosis of COPD who have a history of kidney or liver transplantation.
* People with a diagnosis of COPD who present severity of symptoms and/or respiratory exacerbations categorized in D presenting an mMRC > 2 and CAT > 10 with >1 hospitalization requirements.
* People who are under pharmacological management with erythropoietin (EPO), antibiotics and / or steroids on a chronic basis.
* People with musculoskeletal injuries that limit the execution of the physical training program or that present medical restrictions for the execution of physical exercise.
* People with a diagnosis of COPD who record active smoking.
* People who are participating in research related to medical, pharmacological or physiotherapeutic intervention protocols.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Nuclear concentration of HIF-1 | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Changes in the nuclear concentration of hypoxia-inducible factor (HIF-1) in plasma. For this, an enzyme-linked immunosorbent assay (ELISA) will be executed using specific antibodies to immobilize the study proteins on a plate for their subsequent detection, with chemiluminescence detection.
VEGF protein synthesis. | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Changes in the synthesis of the Vascular Endoletial Growth Factor (VEGF) protein in plasma. For this, an enzyme-linked immunosorbent assay (ELISA) will be executed using specific antibodies to immobilize the study proteins on a plate for their subsequent detection, with chemiluminescence detection.
Synthesis of EPO protein. | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Changes in the synthesis of Erythropoietin (EPO) protein synthesis in plasma. For this, an enzyme-linked immunosorbent assay (ELISA) will be executed using specific antibodies to immobilize the study proteins on a plate for their subsequent detection, with chemiluminescence detection.

SECONDARY OUTCOMES:
Arm Curl Test | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  The total number of times the dominant arm is flexed and extended during 30 seconds.
Chair Stand Test | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  The total number of times the person gets up and sits in the chair for 30 seconds.
6 Minute WalK Test | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Distance traveled by the person be walking on flat ground for 6 minutes
Chair-Sit and Reach Test | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  While sitting, the person will touch the leg that is stretched out with their hands. The distance in cm from the tip of the fingers to the top of the shoe is measured while sitting. If the fingers of the hands do not reach the foot, the distance will be measured in negative values (-) and if the fingers of the hands exceed the foot, the distance will be recorded in positive values (+)
Back Scratch Test | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  They put their hands touching their back "as if it were scratching." The distance between the tips of the middle fingers of the two hands. If the fingers of the hands do not touch, the distance will be measured in negative values (-). If the fingers of the hands overlap, the distance is recorded in positive values (+).
8-Foot up and go Test | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  The person gets up from the chair and walks as fast as possible by a line to surround a cone located 2.44 meters away and must sit again. The time (minutes and seconds) the person spends doing the exercise is measured.
Forced expired volume in the first second (FEV1) | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Volume of air expelled during the first second of maximum expiration, carried out after maximum inspiration. Percentage of air expelled in the first second of expiration.
Functional Vital Capacity (FVC) | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Maximum volume of expired air, with the maximum possible effort, starting from a maximum inspiration. It is expressed as a volume in milliliters.
FEV1/FVC ratio | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Relationship between Forced Expiratory Volume in the first second (FEV1) and Forced Vital Capacity (FVC). It is expressed as a percentage.
Erythrocyte count | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Percentage of reticulocyte volume in a given volume of blood. Reticulocytes / blood volume * microliter.
Medium corpuscular volume (MCV) | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Average size of red blood cells. MCV(fl) = Hematocrit (%) x 10 / Red blood cells (x 10^6/ul)
Mean Corpuscular Hemoglobin (HCM) | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Average hemoglobin content of each red cell. HCM (pg) = Hemoglobin (g/dl) x 10/Red blood cells (x10^6/ul)
Blood hemoglobin (Hb) | 1. Initial measurement (week 0) before the application of the physical exercise program. 2. Final measurement (week 8) after completion of the intervention program.
  Amount of hemoglobin in blood sample expressed in grams per deciliter. Hb = g/dL

CONTACTS AND LOCATIONS:
Overall Officials: Wilder A Villamil-Parra, Therapist, Principal Investigator — Universidad Nacional de Colombia
Locations (1):
- National university of Colombia, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No
At the moment there are no plans to share data, since this process does not have the endorsement of the ethics committee.

REFERENCES:
- [Background] Lee SW, Hwang HH, Hsu PW, Chuang TY, Liu CW, Wu LS. Whole-genome methylation profiling from PBMCs in acute-exacerbation COPD patients with good and poor responses to corticosteroid treatment. Genomics. 2019 Dec;111(6):1381-1386. doi: 10.1016/j.ygeno.2018.09.010. Epub 2018 Sep 21. PMID 30248490
- [Background] To M, Yamamura S, Akashi K, Charron CE, Haruki K, Barnes PJ, Ito K. Defect of adaptation to hypoxia in patients with COPD due to reduction of histone deacetylase 7. Chest. 2012 May;141(5):1233-1242. doi: 10.1378/chest.11-1536. Epub 2011 Dec 15. PMID 22172637
- [Background] Ito K, Ito M, Elliott WM, Cosio B, Caramori G, Kon OM, Barczyk A, Hayashi S, Adcock IM, Hogg JC, Barnes PJ. Decreased histone deacetylase activity in chronic obstructive pulmonary disease. N Engl J Med. 2005 May 12;352(19):1967-76. doi: 10.1056/NEJMoa041892. PMID 15888697
- [Background] Semenza GL. Hypoxia-inducible factor 1 (HIF-1) pathway. Sci STKE. 2007 Oct 9;2007(407):cm8. doi: 10.1126/stke.4072007cm8. PMID 17925579
- [Background] Fu X, Zhang F. Role of the HIF-1 signaling pathway in chronic obstructive pulmonary disease. Exp Ther Med. 2018 Dec;16(6):4553-4561. doi: 10.3892/etm.2018.6785. Epub 2018 Sep 21. PMID 30542404
- [Background] Chen LJ, Xu W, Li YP, Ma LT, Zhang HF, Huang XB, Yu GG, Ma XQ, Chen C, Liu YH, Wu J, Wang LJ, Xu Y. Lycium barbarum Polysaccharide Inhibited Hypoxia-Inducible Factor 1 in COPD Patients. Int J Chron Obstruct Pulmon Dis. 2020 Aug 24;15:1997-2004. doi: 10.2147/COPD.S254172. eCollection 2020. PMID 32921997
- [Background] Kanazawa H, Yoshikawa J. Elevated oxidative stress and reciprocal reduction of vascular endothelial growth factor levels with severity of COPD. Chest. 2005 Nov;128(5):3191-7. doi: 10.1378/chest.128.5.3191. PMID 16304261
- [Result] Tao H, Luo W, Pei H, Zhu S, Zhang M, Chen B, He J, Zhang M, Zhou R. [Expression and significance of hypoxia-inducible factor-1alpha in patients with chronic obstructive pulmonary disease and smokers with normal lung function]. Xi Bao Yu Fen Zi Mian Yi Xue Za Zhi. 2014 Aug;30(8):852-5. Chinese. PMID 25108440
- [Derived] Villamil-Parra W, Cristancho-Mejia E, Ramon Torrella J, Mancera-Soto EM. Effects of a physical exercise program on HIF-1alpha in people with Chronic Obstructive Pulmonary Disease living at high altitude: study protocol for a clinical trial. Trials. 2023 Oct 29;24(1):698. doi: 10.1186/s13063-023-07698-y. PMID 37899477

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT04955977/SAP_000.pdf
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT04955977/ICF_001.pdf